CLINICAL TRIAL: NCT07337369
Title: Cultural Adaptation of Cognitive Behavioral Therapy for Insomnia for the Arab World
Brief Title: Cultural Adaptation of CBTi for the Arab World
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Charles M. Morin, professor at the School of Psychology, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-073
Record Dates: First submitted 2025-12-14; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Insomnia Disorder; Insomnia; Cultural Adaptation
Keywords: culturally tailored CBTi; insomnia; RCT; intercultural intervention; cultural adaptation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial design. Participants are randomly assigned in equal proportions to one of three groups: surface-adapted CBTi, surface- and deep-adapted CBTi, or a wait-list control condition. Groups are followed concurrently, and outcomes are compared between groups across multiple assessment time points.
Who Masked: Participant
Masking Description: Only participants are masked in this study. Participants are unaware of which version of the culturally adapted CBTi they receive or whether they are assigned to an active treatment or the wait-list condition. The therapist and research team are not masked due to the nature of the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wait-list (No Intervention): received treatment (SD-CBTi) after an 8-week wait
- Surface level adaptation to CBTi (Experimental): Therapy was delivered virtually to match participants' preferences and reduce barriers to access. The program was presented as sleep-focused to reduce mental health stigma and included additional psychoeducation about insomnia and available treatments. Engagement and retention were supported through frequent session reminders and access to the research team between sessions. These surface-level adaptations were identical for both intervention groups.
  In the surface-adapted CBTi group, the therapist used a directive approach, and 90-minute sessions equally emphasized cognitive and behavioral techniques.
  Interventions: Behavioral: Surface level adaptation
- Surface+Deep level adaptation to CBTi (Experimental): Delivered in a group format emphasizing collectivist values to reduce loneliness related to insomnia and to involve family support through targeted psychoeducational materials. Session content reflected culturally specific experiences of insomnia, such as racing thoughts and spiritual coping strategies. The first two sessions focused primarily on cognitive techniques, followed by an equal emphasis on cognitive and behavioral strategies from session three onward. Sessions concluded with a brief spiritual mantra practice combining breathing and prayer, and the therapist adopted a less directive approach.
  Deep-level adaptations followed the Cultural Treatment Adaptation Framework and included a culturally grounded explanatory model of insomnia that emphasized culturally relevant causes, symptoms, coping strategies, and help-seeking behaviors. Cultural elements were integrated into sleep hygiene, behavioral, and cognitive techniques, including guidance on prayer, co-sleeping, gradual sle
  Interventions: Behavioral: Surface+deep level adaptations

INTERVENTIONS:
Behavioral: Surface+deep level adaptations — 2levels of deep adaptations. Core-modification. The explanatory model of insomnia for Arabs (El Gewely et al., 2024) replaced the standard "3P model" in session 1, highlighting cultural: causes, symptoms like "Thinking a lot", adaptative strategies (i.e. spiritual mantras) and help-seeking behaviors.
  Core-additions. Additional cultural elements were added to: sleep hygiene, cognitive and behavioral techniques.
  Sleep hygiene. Instructions targeted stimulating sleep environment, co-sleeping practices, prayers, herbal consumptions as well as biphasic sleep culture (e.g. allowing for 20-30 min nap from 3-6PM).
  Behavioral techniques. Sleep restriction was gradual: first two sessions participants were advised to follow regular sleep schedule; from session 3, sleep windows of at least six hours were allocated. Morning prayer practice was considered when needed. Additional hour was given on sleep windows during weekends to accommodate social commitments. Stimulus control included spiritu
  Arms: Surface+Deep level adaptation to CBTi
Behavioral: Surface level adaptation — Engagement. Therapy was offered virtually to accommodate participants' preference over internet-based compared to in-person treatment, based on our cohort and prior research (Ellis & Miller-Graff, 2021). The intervention was framed as a sleep focused program to decrease mental health stigma. Additional psychoeducational increased awareness of insomnia treatment options. To enhance retention, frequent session reminders were sent, and participants were encouraged to contact the research team (MEG and NA) between sessions when needed. These surface-level adaptation were identical for S and SD-CBTi groups.
  Delivery. With S-CBTi group, the therapist was directive. Sessions lasted 90-minutes and incorporated cognitive and behavioral techniques equally.
  Arms: Surface level adaptation to CBTi

SUMMARY:
The goal of this clinical trial is to learn whether culturally adapted versions of Cognitive Behavioral Therapy for insomnia (CBTi) can reduce insomnia severity and improve sleep and mood outcomes in Arab adults with insomnia. The main questions it aims to answer are:

Does culturally adapted CBTi (surface-level or surface + deep-level adaptations) reduce insomnia severity compared to a wait-list control condition?

Are there differences in treatment efficacy between surface-level adaptations and combined surface + deep-level cultural adaptations of CBTi?

Researchers will compare surface-level adapted CBTi, surface + deep-level adapted CBTi, and a wait-list control group to see if culturally adapted CBTi improves insomnia symptoms, sleep parameters, dysfunctional beliefs about sleep, anxiety, depression, and fatigue.

Participants will:

Be randomly assigned to one of three groups: surface-level adapted CBTi, surface + deep-level adapted CBTi, or a wait-list control

Receive a culturally adapted CBTi intervention or remain on a wait-list during the study period

Complete self-report questionnaires assessing insomnia severity, sleep beliefs, mood, and fatigue

Complete sleep diaries at multiple time points across the study duration

DETAILED DESCRIPTION:
Insomnia is a common sleep problem that affects how people fall asleep, stay asleep, and feel during the day. One of the most effective non-medication treatments for insomnia is Cognitive Behavioral Therapy for Insomnia (CBTi). CBTi helps people change unhelpful thoughts and behaviors related to sleep. However, most CBTi programs have been developed and tested in Western countries, and much less is known about how well they work for people from other cultural backgrounds.

Research has shown that individuals from southern cultures, including Arab populations, are often underrepresented in mental health research. This gap is important because culture influences how people understand health problems, seek help, and engage with treatment. Two key findings motivated the current study. First, earlier research found that Syrians showed lower engagement in CBTi, suggesting that standard CBTi may not fully meet the needs of Arab clients. Second, our own qualitative research showed that Arabs often understand sleep and insomnia in culturally specific ways. For example, insomnia is commonly described as a mental or cognitive issue-often referred to as "overthinking"-rather than as a purely biological sleep disorder. Many people also hold social or spiritual explanations for insomnia, such as the belief that sleep problems may be caused by the evil eye or reflect a lack of faith. These beliefs can influence whether and how individuals seek help, with many turning to spiritual practices rather than psychological treatments.

Together, these findings suggest that tailoring CBTi to Arab cultural beliefs and practices may improve its relevance and effectiveness. To guide this process, the study used the Cultural Treatment Adaptation Framework (CTAF), a research-based model that distinguishes between surface-level adaptations, which focus on how treatment is delivered (for example, language, format, and engagement strategies), and deep-level adaptations, which modify core elements of treatment to reflect cultural values, beliefs, and explanatory models of illness.

This pilot randomized controlled trial aimed to compare:

1. A surface-adapted version of CBTi (S-CBTi)
2. A combined surface- and deep-adapted version of CBTi (SD-CBTi)
3. A wait-list control condition (WL)

The main goal was to examine whether culturally adapted CBTi improves insomnia symptoms among Arab adults and whether adding deep-level cultural adaptations provides additional benefits beyond surface-level changes alone.

The study tested two main hypotheses:

1. Both adapted CBTi programs would reduce insomnia severity more than the wait-list condition.
2. The combined surface- and deep-adapted CBTi would lead to greater improvements than the surface-adapted CBTi alone.

The study was a single-blind randomized controlled trial, meaning that participants did not know which version of treatment they were receiving, but the therapist did. Participants were recruited between September 2022 and June 2023 through social media and referrals from a sleep clinic in Cairo, Egypt.

Ethical approval was obtained from the Université Laval Research Ethics Committee, and all participants provided written informed consent before taking part. The study followed internationally recognized guidelines for conducting and reporting clinical trials.

Participants were randomly assigned to one of three groups in equal numbers. An independent statistician ensured that the group assignment process was concealed until all participants had been enrolled. Outcomes were measured at four time points: before treatment began, halfway through treatment, immediately after treatment, and three months later.

Adults aged 18 and older were eligible if they identified as Arab, spoke Arabic, and had parents and grandparents raised in an Arab cultural context, including countries in North Africa, the Middle East, and the Arabian Peninsula. Participants had to meet diagnostic criteria for insomnia and report at least moderate insomnia symptoms. People who worked night shifts, used sleep-altering medications, had certain untreated mental health or sleep disorders, or used cannabis frequently were excluded to ensure participant safety and clarity of results.

Both CBTi programs consisted of six group sessions delivered over eight weeks via videoconference, reflecting participants' preference for online treatment and reducing barriers related to access and stigma. Sessions were conducted in Arabic by a bilingual therapist of Arab origin who was trained in CBTi and intercultural clinical practice. Groups included 5 to 8 participants.

Participants in the wait-list group did not receive treatment during the first eight weeks but were offered the culturally adapted CBTi afterward.

Surface-level adaptations focused on improving engagement and accessibility. The program was presented as a sleep-focused intervention rather than a mental health treatment to reduce stigma. Participants received reminders between sessions and were encouraged to contact the research team for support. Sessions followed standard CBTi principles, with equal emphasis on cognitive and behavioral strategies, and the therapist used a more directive style.

In addition to the surface-level changes described above, the SD-CBTi program incorporated deep cultural adaptations. These adaptations addressed how insomnia is understood and experienced within Arab cultures.

* A culturally relevant explanation of insomnia that emphasized overthinking, social stressors, and spiritual meanings, rather than relying solely on Western biomedical models.
* Integration of collectivist values through group discussion, shared experiences, and educational materials designed for family members.
* Adaptations to sleep hygiene recommendations that considered co-sleeping, prayer practices, herbal remedies, and common sleep patterns such as daytime napping.
* Gradual sleep restriction and flexible scheduling to accommodate religious practices, social obligations, and weekends.
* Cognitive strategies that directly addressed culturally shaped beliefs, such as the idea that insomnia reflects weak faith.
* Inclusion of spiritual practices, such as brief breathing exercises followed by prayer, at the end of sessions.
* Discussion of culturally relevant situations that may disrupt sleep, including Ramadan, seasonal changes, and family responsibilities.

The therapist adopted a less directive, more collaborative style in this condition, and sessions were slightly longer to allow space for discussion and reflection.

The primary outcome was insomnia severity, measured using a validated Arabic version of the Insomnia Severity Index (ISI). Improvements were considered clinically meaningful if participants showed a substantial reduction in symptoms or no longer met criteria for insomnia.

Secondary outcomes included:

* Beliefs and attitudes about sleep
* Anxiety and depression symptoms
* Fatigue
* Objective sleep patterns reported in daily sleep diaries, such as time to fall asleep and total sleep time

These measures allowed researchers to examine not only whether sleep improved, but also whether participants felt better emotionally and functioned better during the day.

The study used statistical methods that included all participants as originally assigned, even if they did not complete every assessment. This approach reflects real-world treatment conditions. Analyses compared changes over time between the three groups and examined whether improvements were maintained at the three-month follow-up.

This study addresses an important gap in sleep and mental health research by focusing on Arab populations, who are often overlooked in clinical trials. By systematically testing cultural adaptations to CBTi, the study helps clarify whether and how evidence-based treatments can be tailored for different cultural contexts. The findings have the potential to inform more inclusive, culturally responsive sleep interventions and improve access to effective insomnia treatment for Arab communities worldwide.

ELIGIBILITY:
Inclusion Criteria:

* 18 + years
* Arab descent (parents and grandparents born and raised in an Arab culture (Egypt, Morrocco, Algeria, Tunisia, Palestine, Libya, Sudan, Lebanon, Syria, Saudi Arabic, Yemen, UAE, Oman, Kuwait, Qatar, Bahrain))
* Arabic speaking
* if migrated, after the age of 12
* meeting DSM-5 insomnia diagnosis, assessed by Insomnia Diagnostic Interview (Morin & Espie, 2003)
* ISI score > 10
* no prior CBTi
* stable medication or no psychiatric disorder as assessed by MINI Psychiatric Interview (Sheehan et al., 1998).

Exclusion Criteria:

* night-shift or atypical schedule (bedtime after 3am, wake up after 11 am, >2 nights/week)
* sleep altering medications
* untreated comorbidity requiring imminent intervention as evaluated by MINI (Sheehan et al., 1998)
* psychotic or bipolar disorder
* other sleep disorder
* cannabis use > 2 days/week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2023-12-23 (Actual)

PRIMARY OUTCOMES:
Insomnia severity index | pre-treatment, mid-treatment (6 weeks after time 1), post-treatment (approximately 9 weeks after time 1) and 3 months follow-up (approximately 3 months after post-treatment)
  The primary outcome was the Arabic validated version of the ISI. This scale shows strong internal consistency (Cronbach's alpha = .84) and convergent validity, correlating with the Pittsburgh Sleep Quality Index among Arabs (Suleiman & Yates, 2011). The ISI is a 7-item self-reported measure of night-time and daytime insomnia symptoms (Bastien et al., 2001). Each item is rated on a five-point Likert scale (0-4). ISI scores range from 0-28, with higher scores indicating severe symptoms (Bastien et al., 2001; Morin et al., 2011). Since ISI score interpretation has not been yet validated for Arabs. ISI scores were interpreted based on Bastien et al. (2001) guidelines: non-clinical (0-7), subthreshold insomnia (8-14), clinical insomnia (moderate (15-21) and severe severity (22-28).

SECONDARY OUTCOMES:
Hospital Anxiety and Depression scale | baseline (time 1) and post-treatment (approximately 9 weeks after time 1)
  HADS includes 14 items assessing anxiety and depression, rated on a 4-point scale (Cronbach's alpha: .83 and .77 respectively) (Terkawi et al., 2017). Since score interpretation for Arabs is lacking, they were interpreted per Zigmond & Snaith (1983): subclinical (0-7), borderline case (8-10), and clinically significant anxiety or depression (11-21).
Multidimensional Fatigue Inventory | baseline (time 1) and post-treatment (approximately 9 weeks after time 1)
  MFI includes 20 items rated on a Likert scale, with higher scores indicating greater fatigue (Smets et al., 1995). It evaluates five factors: general, physical and mental fatigue, reduced motivation and activity (Cronbach's alphas ranging from .12 to .66) (Haggag & Soliman, 1997).
Dysfunctional Beliefs and Attitudes about sleep | baseline (time 1), post-treatment (approximately 9 weeks after time 1) and at 3-month follow-up (approximately 3 months after post-treatment ((approximately 3 months after post-treatment))
  DBAS-16 captures frequent maladaptive beliefs and attitudes about sleep (Morin et al., 2007). This scale was translated to Arabic by our research team. DBAS-16 is composed of four factors: consequences (Factor 1), worry/helplessness (Factor 2), expectations (Factor 3) and medication use (Factor 4) (Morin et al., 2007). Items are scored 0-10, with the total average score from 0-10.. Cronbach alpha was .77 for clinical samples (Morin et al., 2007).
Sleep diary | baseline (time 1), post-treatment (approximately 9 weeks after time 1) and at 3-month follow-up (approximately 3 months after post-treatment)
  Sleep measures (i.e. sleep onset latency, wake after sleep, total sleep, time in bed, sleep efficiency) were collected using the consensus sleep diary (Carney et al., 2012).

CONTACTS AND LOCATIONS:
Locations (1):
- Neuromed Clinic, Laval, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El Gewely, M., Leanza, Y., Moustafa, R. R., Attia, N., Hesham, H., Bastien, C., & Morin, C. M. (2024). Explanatory model of sleep and insomnia in the Arab world: A qualitative study. Sleep Medicine, 115, S176-S177. https://doi.org/10.1016/j.sleep.2023.11.500
- [Background] Zhou ES, Ritterband LM, Bethea TN, Robles YP, Heeren TC, Rosenberg L. Effect of Culturally Tailored, Internet-Delivered Cognitive Behavioral Therapy for Insomnia in Black Women: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Jun 1;79(6):538-549. doi: 10.1001/jamapsychiatry.2022.0653. PMID 35442432